CLINICAL TRIAL: NCT01143025
Title: Peritoneal Nebulization of Ropivacaine for Postoperative Pain Control After Laparoscopic Cholecystectomy
Brief Title: Intraperitoneal Ropivacaine Nebulization for Pain Control After Laparoscopic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: San Gerardo Hospital (Other)
Collaborators: University of Milano Bicocca (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Azienda L'ULSS 15 Alta Padovana (Other); Gruppo Ospedaliero San Donato, Policlinico San Pietro, Ponte San Pietro, Bergamo (Unknown); Azienda U.S.L. della Valle d'Aosta, Ospedale Regionale Umberto Parini (Unknown)
Responsible Party: Pablo M Ingelmo, MD, First Service of anesthesia and intensive care. San Gerardo Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR HSG 01 2010
Record Dates: First submitted 2010-06-09; First posted 2010-06-14 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Laparoscopic Cholecystectomy; Nebulization; Ropivacaine
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ropivacaine 50 mg (Active Comparator): Preoperative nebulization of 50 mg of Ropivacaine in the peritoneal cavity
  Interventions: Drug: Ropivacaine 50 mg
- Ropivacaine 100 mg (Experimental): Preoperative nebulization of 100 mg of Ropivacaine in the peritoneal cavity
  Interventions: Drug: Ropivacaine 100 mg
- Ropivacaine 150 mg (Experimental): Preoperative nebulization of 150 mg of Ropivacaine in the peritoneal cavity
  Interventions: Drug: Ropivacaine 150 mg

INTERVENTIONS:
Drug: Ropivacaine 50 mg — Preoperative nebulization of 50 mg of Ropivacaine in the peritoneal cavity
  Other Names: Nebulization; Ropivacaine
  Arms: Ropivacaine 50 mg
Drug: Ropivacaine 100 mg — Preoperative nebulization of 100 mg of Ropivacaine in the peritoneal cavity
  Other Names: Nebulization; Ropivacaine
  Arms: Ropivacaine 100 mg
Drug: Ropivacaine 150 mg — Preoperative nebulization of 150 mg of Ropivacaine in the peritoneal cavity
  Other Names: Nebulization; Ropivacaine
  Arms: Ropivacaine 150 mg

SUMMARY:
The purpose of this study is to assess if intraperitoneal nebulization of Ropivacaine 50 mg, 100 mg or 150 mg may prevent the use of morphine during the first day after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Intraperitoneal aerosolization of Bupivacaine 50 mg after laparoscopic cholecystectomy has been proved to significantly reduce postoperative pain, morphine consumption and incidence of postoperative nausea and vomiting in comparison with patients receiving direct instillation of Bupivacaine 50 mg or placebo.

Ropivacaine can be effectively administrated with non-heating nebulizers (AeronebPro®). In a recent study our group found that nebulization of Ropivacaine 30 mg with the AeronebPro® before or after laparoscopic cholecystectomy significantly reduced postoperative pain and morphine consumption. Nonetheless, most patients still need strong opioid based analgesia after surgery.

We hypothesize that intraperitoneal nebulization of Ropivacaine 100 mg and 150 mg (maximum recommended dose in adults 300 mg or up to 3 mg/kg) may prevent the use of morphine during the first day after surgery maintaining ropivacaine plasma levels below toxic concentration.

ELIGIBILITY:
Inclusion Criteria:

* Females and Males 18-75 years old
* ASA Score I-III
* Scheduled for laparoscopic cholecystectomy
* Free from pain in preoperative period
* Not using analgesic drugs before surgery
* Without cognitive impairment or mental retardation
* Written informed consent

Exclusion Criteria:

* Emergency/urgency surgery
* Postoperative admission in an intensive care unit
* Cognitive impairment or mental retardation
* Progressive degenerative diseases of the CNS
* Seizures or chronic therapy with antiepileptic drugs
* Severe hepatic or renal impairment
* Pregnancy or lactation
* Allergy to one of the specific drugs under study
* Acute infection or inflammatory chronic disease
* Alcohol or drug addiction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Morphine consumption (mg) | Up to 48 hours
  The total dose of morphine at every evaluation after awakening will be quantified using the PACU clinical chart and/or PCA infusers memory display

SECONDARY OUTCOMES:
Ropivacaine pharmacokinetics profile: Plasma Concentration of Ropivacaine | Up to 360 minutes
  We will perform a pharmacokinetic analysis through venous samples collected at 20, 40, 60, 90, 240, and 360 minutes after the end of nebulization.
Ropivacaine pharmacokinetics profile: Tissue drug analysis | Up to 2 hours
  Tissue samples (at least 2 g of tissue) from parietal peritoneum will be taken at the end of surgery . The supernatant will be analised with mass-spectrometry
Postoperative Pain | Up to 48 hours
  Postoperative pain will be assessed by numeric ranking scale (NRS 0 to 10 points) at rest (static NRS) and after a deep inspiration or cough (dynamic NRS). Pain after surgery will be differentiated as abdominal, wall pain, port wound pain and/or shoulder pain. The proportion of patients with adequate pain control after surgery (dynamic NRS < 3) will also be assessed.
Time of unassisted walking | Up to 48 hours
  Unassisted walking time is defined as the time in hours between PACU discharge and when the patient is able to walk out of his room and back to bed without any assistance.
Hospital morbidity | Up to 48 hours
  All complications or adverse effects associated or possibly associated with the interventions under study, surgery or anesthesia will be quantified using the anesthesia charts, surgical charts, surgical database.
Time and condition for hospital discharge | Up to 48 hours
  We define hospital stay as the elapsed time between surgery and hospital discharge, in days. We also evaluate the hospital stay with the post-anesthetic discharge scoring system (Modified-PADSS).
Quality of life after surgery | Four weeks after surgery
  Quality of life will be assessed using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Allegri, MD, Study Chair — Servizio Anestesia e Rianimazione I e Terapia del Dolore, Fondazione IRCCS Policlinico San Matteo, Pavia; Mario Regazzi, MD, Study Chair — Head of Clinical PK and TDM Laboratory, Foundation IRCCS Policlinico San Matteo, Pavia; Ernesto Pizzirani, MD, Study Chair — U.O.C. Anestesia e Rianimazione. A.O. U.L.S.S.15 "Alta Padovana", Presidio Camposampiero. Camposampiero - Padova; Fiorenza Franceschi, MD, Study Chair — U.O.C. Anestesia e Rianimazione. A.O. U.L.S.S.15 "Alta Padovana", Presidio Camposampiero. Camposampiero - Padova; Armando Alborghetti, MD, Study Chair — U.O.C. Anestesia e Rianimazione. Ospedale di Ponte San Pietro. Bergamo; Alessandro Albani, MD, Study Chair — U.O. Anestesia e Rianimazione. Ospedale Regionale "U. Parini", Aosta; Pierre Diemusch, MD, Study Chair — Servizio di Anestesia e rianimazione chirurgica. Hospital de Hautepierre. Università di Strasburgo.
Locations (1):
- San Gerardo Hospital, Monza, MB, Italy

REFERENCES:
- [Background] Greib N, Schlotterbeck H, Dow WA, Joshi GP, Geny B, Diemunsch PA. An evaluation of gas humidifying devices as a means of intraperitoneal local anesthetic administration for laparoscopic surgery. Anesth Analg. 2008 Aug;107(2):549-51. doi: 10.1213/ane.0b013e318176fa1c. PMID 18633034
- [Background] Schlotterbeck H, Schaeffer R, Dow WA, Diemunsch P. Cold nebulization used to prevent heat loss during laparoscopic surgery: an experimental study in pigs. Surg Endosc. 2008 Dec;22(12):2616-20. doi: 10.1007/s00464-008-9841-z. Epub 2008 Mar 18. PMID 18347861
- [Result] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268